CLINICAL TRIAL: NCT02269189
Title: A Randomized, Double-blind Within Dose, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Repeated Oral Doses (15-day Dosing) of BIIL 284 BS in Adult (300 mg) and Pediatric (150 mg) Cystic Fibrosis Patients
Brief Title: Safety, Tolerability and Pharmacokinetics of BIIL 284 BS in Adult and Pediatric Cystic Fibrosis (CF) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.37
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — amelubant

ARMS (3):
- BIIL 284 BS, high dose in adult patients (Experimental)
  Interventions: Drug: BIIL 284 BS, high dose
- BIIL 284 BS, low dose in pediatric patients (Experimental)
  Interventions: Drug: BIIL 284 BS, low dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 BS, high dose
  Arms: BIIL 284 BS, high dose in adult patients
Drug: BIIL 284 BS, low dose
  Arms: BIIL 284 BS, low dose in pediatric patients
Drug: Placebo
  Arms: Placebo

SUMMARY:
Safety, tolerability and pharmacokinetics following repeated doses (15-day dosing)

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 6 years (pediatric 6 - 17 years inclusive; adult ≥ 18 years); minimum weight requirement of 20 kg
* Confirmed diagnosis of CF (positive sweat chloride ≥ 60 milliequivalents (mEq)/liter (by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations consistent with CF accompanied by one or more clinical features with the CF phenotype
* Forced expiratory volume in one second (FEV1) > 25% predicted (using prediction equation's of Knudson et al)
* Clinically stable with no evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within 2 weeks of screening
* Females of child bearing potential must have a negative pregnancy test at screening and, if sexually active, must be willing to use a double-barrier form of contraception for the duration of the study
* The patient or the patient's legally acceptable representative must be able to give informed consent in accordance with International Conference on Harmonization (ICH) Good Clinical Practice (GCP) guidelines and local legislation
* The patient must be able to swallow the BIIL 284 tablet whole
* Patients taking a chronic medication must be willing to continue this therapy for the entire duration of the study

Exclusion Criteria:

* Patients with a history of allergy/hypersensitivity (including medication allergy) which is deemed relevant to the trial as judged by the Investigator
* Patients who have participated in another study with an investigational drug (including BI Trial 543.36) within one month or 6 half-lives (whichever is greater) preceding the screening visit
* Patients with known substance abuse, including alcohol or drug abuse, within 30 days prior to screening
* Female patients who are pregnant or lactating
* Patients who are unable to comply with breakfast requirements prior to dosing
* Patients who have received IV, oral or inhaled antibiotics or corticosteroids for a pulmonary exacerbation within 2 weeks of screening
* Patients who have started a new chronic medication for CF within 2 weeks of screening
* Patients with documented persistent colonization with B. cepacia (defined as more than one positive culture within the past year)
* Patients with clinically significant findings on chest x-ray which in the opinion of the Investigator precludes the patient's participation in the trial
* Patients with oxyhemoglobin saturation in room air < 90% by pulse oximetry
* Patients with hemoglobin < 9.0 g/dL; platelets < 100x10**9/L; prothrombin time (PT) > 1.5 times the upper limit of normal, serum glutamic-oxaloacetic transaminase (ALT) or serum glutamic-pyruvic transaminase (AST) > 2 times the upper limit of normal; creatinine > 1.8 mg/dL (adults) or > 1.4 mg/dL (pediatrics) at screening
* Clinically significant disease or medical condition other than CF or CF-related conditions that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. This includes significant hematological, hepatic, renal, cardiovascular, and neurologic disease. Patients with diabetes may participate if their disease is under good control prior to screening.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-04; Primary Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in physical examination | Pre-dose and 72 hours after last drug administration
Number of patients with clinically relevant findings in vital signs | Up to 72 hours after last drug administration
  blood pressure, pulse rate, respiratory rate, body temperature
Number of patients with clinically relevant changes in spirometry | Pre-dose, up to 72 hours after last drug administration
Number of patients with clinically relevant changes in oximetry | Pre-dose, up to 72 hours after last drug administration
Number of patients with clinically relevant changes in 12-lead ECG | Pre-dose, up to 72 hours after last drug administration
Number of patients with clinically relevant findings in laboratory evaluation | Up to 72 hours after last drug administration
Number of patients with adverse events | Up to 72 hours after last drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma (AUC) | Up to 72 hours after last drug administration
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 72 hours after last drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | Up to 72 hours after last drug administration
Concentration of the analyte in plasma after 24 hours (C24h) | 24 hours after drug administration
Pre-dose concentration of the analyte in plasma immediately before administration of the next dose (Cpre) | Up to day 16
Terminal rate constant of the analyte in plasma (λz) | Up to 72 hours after last drug administration
Terminal half-life of the analyte in plasma (t1/2) | Up to 72 hours after last drug administration
Mean residence time of the analyte in the body at steady state (MRTss) | Up to 72 hours after last drug administration
Apparent volume of distribution during the terminal phase λz following extravascular administration at steady state (Vz,ss/F) | Up to 72 hours after last drug administration
Accumulation ratio for AUC after the 15th dose over the dosing interval compared to the first dose (RA,AUC) | day 1, day 15
Accumulation ratio for Cmax after the 15th dose over the dosing interval compared to the first dose (RA,Cmax) | day 1, day 15